CLINICAL TRIAL: NCT06370949
Title: Comparison of the Effectiveness of Bupivacaine and Bupivacaine+Dexmedetomidine Combination in Transversus Abdominis Plane* Block in Colorectal Cancer Surgery
Brief Title: The Effectiveness of Bupivacaine and Bupivacaine+Dexmedetomidine Combination in Transversus Abdominis Plane* Block
Acronym: TAP
Status: Not yet recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Beyza Seker, Resident Anaesthesiologist, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2024-01/17
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: colorectal cancer; colorectal cancer surgery; colorectal neoplasym; transversus abdominis plane; transversus abdominis plane block
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bupivacaine: Ultrasonography (USG) guided bilateral TAP block:20 ml %0,25 concentration bupivacain
  Interventions: Drug: Bupivacain
- bupivacaine+dexmedetomidine: Ultrasonography (USG) guided bilateral TAP block: 20 ml %0,25 concentration bupivacain+ 0.5 mcg/kg dexmedetomidine
  Interventions: Drug: bupivacain+dexmedetomidine

INTERVENTIONS:
Drug: Bupivacain — Ultrasonography (USG) guided bilateralTAP block:20 ml %0,25 concentration bupivacain
  Groups: bupivacaine
Drug: bupivacain+dexmedetomidine — Ultrasonography (USG) guided bilateral TAP block: 20 ml %0,25 concentration bupivacain+ 0.5 mcg/kg dexmedetomidine
  Groups: bupivacaine+dexmedetomidine

SUMMARY:
Transversus abdominis plane (TAP) block is an anesthesia method that provides somatic analgesia to the anterior and lateral abdominal walls. Thus, TAP block is widely implemented in perioperative management of colorectal cancer patients.

Researchers aimed to evaluate the analgesic effectiveness and duration of effect of dexmedetomidine added to bupivacaine in the TAP block applied in colorectal cancer surgeries.

DETAILED DESCRIPTION:
Transversus abdominis plane (TAP) block is an anesthesia method that provides somatic analgesia to the anterior and lateral abdominal walls. With the increasing use of ultrasound guidance during peripheral nerve blocks, trunk blocks such as the transversus abdominis plane (TAP) block are widely used for analgesia after abdominal surgery.

The advantages of TAP block include being less invasive than epidural analgesia, lower incidence of hypotension, and shorter hospital stay. Due to these advantages, TAP block has become a widely preferred method.

Researchers aimed to evaluate the analgesic effectiveness and duration of effect of dexmedetomidine added to bupivacaine in the TAP block applied in colorectal cancer surgeries. The study will be conducted in a tertiary oncology hospital in Turkey and 84 colorectal cancer patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer diagnosis
* undergoing colorectal cancer surgery

Exclusion Criteria:

* allergic reaction to local anesthetics
* bleeding anomalies
* infection in TAP block area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will evaluate colorectal cancer patients from Ankara Dr. Abdurrahman Yurtaslan Oncology Train and Research Hospital who will undergo colorectal cancer surgery.
  The investigators will exclude patients who no longer want to participate at any part of the trial.
  A total of 84 patients' data will be collected.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Analgesic effectiveness of bupivacain and bupivacain+dexmedetomidine combination in colorectal cancer surgery | postoperative day two
  Numeric Rating Scales of two groups in postoperative period. The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

CONTACTS AND LOCATIONS:
Overall Officials: Beyza Seker, MD, Principal Investigator — Resident MD
Locations (1):
- Turkey Dr.Abdurrahman Yurtaslan Ankara Oncology Train and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)